

# Statistical Analysis Plan for CLA306-P001 / NCT04908488 Title: Clinical Performance of Two Daily Disposable Toric Soft Contact Lenses



This version of the Statistical Analysis Plan is based on Version 2.0 of the study protocol.

#### **Executive Summary:**

Key Objectives:

The primary objective of this study is to demonstrate noninferiority in the visual acuity (VA) at distance when wearing PRECISION1<sup>TM</sup> for Astigmatism (P1fA) contact lenses compared to 1-DAY ACUVUE<sup>®</sup> MOIST for ASTIGMATISM (AMfA) contact lenses.

Decision Criteria for Study Success:

Success of this study will be based on demonstration of noninferiority in distance VA with P1fA when compared to AMfA, using a margin of 0.05.

# **Table of Contents**

| Sta | atistical A | Analysis Plan for CLA306-P001 | 1 |
|---|---|---|---|
| Ta | ble of Cor | ontents | 3 |
| Lis | st of Table | es | 4 |
| Lis | st of Figur | ıres | 4 |
| 1 | STUDY | Y OBJECTIVES AND DESIGN | 5 |
| | 1.1 | Study Objectives | 5 |
| | 1.2 | Study Description | |
| | 1.3 | Randomization | 6 |
| | 1.4 | Masking | 7 |
| | 1.5 | Interim Analysis | 7 |
| 2 | ANALY | YSIS SETS | 7 |
| | 2.1 | Safety Analysis Sets | 7 |
| | 2.2 | Full Analysis Set | |
| 3 | SUBJEC | CT CHARACTERISTICS AND STUDY CONDUCT SUMMARIE | ES8 |
| 4 | EFFEC7 | TIVENESS ANALYSIS STRATEGY | 8 |
| | 4.1 | Effectiveness Endpoints | 9 |
| | 4.2 | Effectiveness Hypotheses | 10 |
| | 4.3 | Statistical Methods for Effectiveness Analyses | 11 |
| | | 4.3.1 Primary Effectiveness Analysis | 11 |
| _ | | NA ANALYZOIG GER ATTECNA | 1.5 |
| 5 | | Y ANALYSIS STRATEGY | _ |
| | 5.1 | Safety Endpoints | |
| | 5.2 | Safety Hypotheses | |
| | 5.3 | Statistical Methods for Safety Analyses | |
| | 5.4 | Adverse Events | |
| | | 5.4.1 Biomicroscopy Findings/Slit Lamp Examination 5.4.2 Device Deficiencies | |
| | | J. 1.2 DOVICE DEHICION | 1 / |

| 6 | ANALYS | IS STRATEGY FOR OTHER ENDPOINTS1 |
|---|---|---|
| 7 | SAMPLE | SIZE AND POWER CALCULATIONS |
| 8 | REFERENCES18 | |
| 9 | REVISIO | N HISTORY1 |
| 10 | APPENDI | IX1 |
| | | List of Tables |
| Tab | le 1-1 | Study Description Summary |
| Tab | le 10-1 | Schedule of Study Procedures and Assessments |
| E. | 1 1 | List of Figures |
| Figi | ure 1–1 | Flowchart of Study Visits |

#### 1 STUDY OBJECTIVES AND DESIGN

# 1.1 Study Objectives

#### PRIMARY OBJECTIVE(S)

The primary objective of this study is to demonstrate noninferiority in the VA at distance when wearing P1fA contact lenses compared to AMfA contact lenses.



# 1.2 Study Description

Key components of the study are summarized in Table 1-1.

Table 1-1 Study Description Summary

| Study Design | Prospective, randomized, controlled, double-masked, bilateral crossover |
|---|---|
| Study Population | Volunteer subjects aged 18 or over who are habitual toric soft |
| | contact lens wearers (excluding current/previous P1fA and |
| | AMfA contact lens habitual wearers), have at least 3 months of |
| | contact lens wearing experience, and who wear their habitual |
| | lenses at least 5 days per week and at least 10 hours per day. |
| | Target to complete: 100; Planned to enroll: ~110 |
| Number of Sites | ~8 |
| | US |
| Test Product | PRECISION1 <sup>TM</sup> for Astigmatism contact lenses (P1fA), |
| Control Product | 1-DAY ACUVUE® MOIST for ASTIGMATISM (AMfA), |
| Planned Duration of | ~ 22 days total (test and controls): |
| Exposure | Test Product: 8 -0/+3 days |
| | Control Product: 8 -0/+3 days |

| Status: Approved, | Version: 1.0 |
|-------------------|--------------|
| Approved Date: 0 | 7 Jun 2021 |

Document ID: V-CLN-0010097

| Visits | Visit 1 – Screening/Trial Lens Fitting and Evaluation |
|--------|-----------------------------------------------------------------|
| | Visit 2 – Baseline/Dispense Lens 1 (4 -2/+2 days after Visit 1) |
| | Visit 3 – Week 1 Follow-up Lens 1/Dispense Lens 2 (8 -0/+3 |
| | days after Visit 2) |
| | Visit 4 – Week 1 Follow-up Lens 2/Exit (8 -0/+3 days after |
| | Visit 3) |

A study design schematic is depicted in Figure 1–1.

Figure 1–1 Flowchart of Study Visits



#### 1.3 Randomization

A member of the Randomization Programming group at Alcon who is not part of the study team will generate the randomized allocation schedule(s) for lens sequence assignment. Randomization will be implemented in the Electronic Data Capture (EDC)/randomization integration system.

Subjects will be randomized in a 1:1 ratio to receive treatment (lens) in crossover sequence as follows:

| Sequence | EDC/randomization integration system | Lens Name |
|------------|--------------------------------------|-----------|
| Sequence 1 | | P1fA/AMfA |
| Sequence 2 | | AMfA/P1fA |

## 1.4 Masking

This study is double-masked.

#### 1.5 Interim Analysis

There are no plans to conduct an interim analysis and no criteria by which the study would be terminated early based upon statistical determination.

#### 2 ANALYSIS SETS

# 2.1 Safety Analysis Sets

Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. As such, the safety analysis set will include all subjects/eyes exposed to any study lenses evaluated in this study,

For treatmentemergent safety analyses, subjects/eyes will be categorized under the actual study lenses exposed in the corresponding lens sequence.

Adverse events occurring from the time of informed consent but prior to first exposure to study lenses will be summarized in subject listings.

# 2.2 Full Analysis Set

The full analysis set (FAS) is the set of all randomized subjects who are exposed to any study lenses evaluated in this study,



# 3 SUBJECT CHARACTERISTICS AND STUDY CONDUCT SUMMARIES

The following tables will be presented:

- Subject Disposition by Lens Sequence
- Analysis Sets by Lens
- Analysis Sets by Lens Sequence
- Subject Accounting by Lens Sequence
- Demographics Characteristics by Lens Sequence
- Baseline Characteristics by Lens Sequence [lens brand, lens power: sphere, cylinder, axis]

Subject accounting and demographics characteristics tables will be summarized on the safety, full, analysis datasets. Baseline characteristics will be summarized on the full analysis datasets.

In addition, the following subject listings will be provided:

- Listing of Subjects Excluded from Protocol Defined Analysis Sets
- Listing of Lens Sequence Assignment by Investigator
- Listing of Subjects Discontinued from Study

#### 4 EFFECTIVENESS ANALYSIS STRATEGY

| This study defines 1 primary, | effectiveness |
|-------------------------------|---------------|
| endpoint | |

Continuous variables will be summarized using the number of observations, mean, standard deviation, median, minimum, and maximum, as well as confidence intervals (CI) or

confidence limits (CL) where applicable. Categorical variables will be summarized with frequencies and percentages from each category.

All data obtained in evaluable subjects/eyes will be included in the analysis. No imputation for missing values will be carried out

A listing of select effectiveness data will also be provided.

## 4.1 Effectiveness Endpoints

#### **Primary Effectiveness Endpoint**

The primary endpoint is distance VA with study lenses, collected for each eye in logMAR.





# **4.2** Effectiveness Hypotheses

#### **Primary Effectiveness**

The null and alternative hypotheses are formulated in terms of the predefined margin of 0.05 for noninferiority:

$$\begin{split} &H_0 \colon \mu_{(T)} - \mu_{(C)} \ge 0.05 \\ &H_a \colon \mu_{(T)} - \mu_{(C)} \le 0.05 \end{split}$$

where  $\mu_{(T)}$  and  $\mu_{(C)}$  denote the mean distance VA for P1fA and AMfA, respectively, on the logMAR scale.



# 4.3 Statistical Methods for Effectiveness Analyses

# 4.3.1 Primary Effectiveness Analysis

A mixed effects repeated measures model will be utilized to test these hypotheses. The model will include terms for lens, visit, and lens by visit interaction, period, and sequence. Withinsubject correlation due to eye and the crossover design will also be accounted for in the model. Lens difference (P1fA minus AMfA) and the corresponding one-sided 95% upper confidence limit will be computed at Week 1. Noninferiority in distance VA will be declared if upper confidence limit is less than 0.05.







#### 5 SAFETY ANALYSIS STRATEGY

The focus of the safety analysis will be a comprehensive descriptive assessment of occurrence of adverse events as well as the other listed parameters. Therefore, no inferential testing will be done for the safety analysis.

#### 5.1 Safety Endpoints

The safety endpoints are

- Adverse events (AE)
- Biomicroscopy Findings/Slit Lamp Examinations
  - o Limbal hyperemia
  - Bulbar hyperemia
  - Corneal staining
  - Conjunctival staining
  - o Palpebral conjunctival observations
  - o Corneal epithelial edema
  - o Corneal stromal edema
  - Corneal vascularization
  - o Conjunctival compression/indention
  - o Chemosis
  - Corneal infiltrates
  - Other findings
- Device deficiencies

# 5.2 Safety Hypotheses

There are no formal safety hypotheses in this study. The focus of the safety analysis will be a comprehensive descriptive assessment of safety endpoints listed in Section 5.1.

# 5.3 Statistical Methods for Safety Analyses

The analysis set for all safety analyses is defined in Section 2.1. Baseline will be defined as the last measurement prior to exposure to study lenses. Safety variables will be summarized descriptively.

#### **5.4** Adverse Events

The applicable definition of an AE is in the study protocol. All AEs occurring from when a subject signs informed consent to the time of their study exit will be accounted for in the reporting.

Pre-treatment AEs will be separated from treatment-emergent AEs occurring during the study period. A pre-treatment AE is an event that occurs after signing informed consent but prior to exposure to study lens. The period for treatment-emergent AE analysis starts from exposure to study lenses until the subject completes or is discontinued from the study. Each AE will be summarized under the exposed lens based upon the event onset date/time, up until the start of the next lens in the crossover sequence.

The following tables and supportive listings will be provided:

- Incidence of All Ocular Treatment-Emergent Adverse Events
- Incidence of Ocular Serious Treatment-Emergent Adverse Events
- Incidence of All Nonocular Treatment-Emergent Adverse Events
- Incidence of Nonocular Serious Treatment-Emergent Adverse Events
- Listing of All Ocular Treatment-Emergent Adverse Events
- Listing of All Nonocular Treatment-Emergent Adverse Events
- Listing of All Ocular Pre-Treatment Adverse Events
- Listing of All Nonocular Pre-Treatment Adverse Events

# 5.4.1 Biomicroscopy Findings/Slit Lamp Examination

The following tables and supportive listings will be provided:

- Frequency and Percentage for Biomicroscopy Findings by Visit
- Incidence of Increased Severity by 2 or More Grades in Biomicroscopy Findings
- Listing of Subjects With Other Biomicroscopy Findings
- Listing of Subjects With Conjunctival Compression/Indentation or Chemosis
- Listing of Subjects With Increased Severity by 2 or More Grades in Biomicroscopy Findings [This listing will include all relevant visit within the crossover period]
- Listing of Subjects with Infiltrates

#### **5.4.2** Device Deficiencies

The following tables and supportive listings will be provided:

- Frequency of Treatment-Emergent Device Deficiencies
- Listing of Treatment-Emergent Device Deficiencies
- Listing of Device Deficiencies Prior To Treatment Exposure

#### 6 ANALYSIS STRATEGY FOR OTHER ENDPOINTS

Not Applicable.

#### 7 SAMPLE SIZE AND POWER CALCULATIONS

Sample size calculation is based on a prior clinical study which evaluated performance of P1fA and AMfA.

#### **Primary Effectiveness**

To demonstrate noninferiority (margin = 0.05 in logMAR; ½ line in Snellen) in distance VA as a one-tailed hypothesis with  $\alpha$ =0.05, and using a standard deviation of 0.0629 for paired differences, 80% power can be attained with a sample size of 12 (6 per sequence).





#### 8 REFERENCES

Not Applicable.

#### 9 REVISION HISTORY

This is the original (Version 1.0) Statistical Analysis Plan for this study. This version of the Statistical Analysis Plan is based on Version 2.0 of the study protocol.

#### 10 APPENDIX

 Table 10-1
 Schedule of Study Procedures and Assessments

| Procedure / Assessment | Visit 1 Screening / Trial Lens Fitting and Evaluation | Visit 2 Baseline / Dispense Lens 1 | Visit 3 Week 1 Follow-up Lens 1 / Dispense Lens 2 | Visit 4 Week 1 Follow-up Lens 2 / Exit | Unscheduled<br>Visit | Early<br>Exit |
|---|---|---|---|---|---|---|
| | | 4 -2/+2 days after Visit 1 | 8 -0/+3 days after Visit 2 | 8 -0/+3 days after Visit 3 | N/A | N/A |
| Informed Consent | X | - | - | - | - | - |
| Demographics | X | - | - | - | - | - |
| Medical History ∞ | X | X | X | X | (X) | X |
| Concomitant Medications ∞ | X | X | X | X | (X) | X |
| Inclusion / Exclusion | X | - | - | - | - | - |
| Habitual lens information (brand, power) | X | - | - | - | - | - |
| VA with habitual contact lens<br>correction (OD, OS, LogMAR<br>distance)* | X | - | - | X | - | X |
| Keratometry* | X | - | - | - | - | - |
| Manifest refraction* (OD, OS; sphere, cylinder, axis) | X | - | (X) | (X) | (X) | X |
| BCVA* (OD, OS logMAR distance with Manifest refraction) | X | - | (X) | (X) | (X) | X |
| Biomicroscopy | X | X | X | X | (X) | X |
| Trial lens fitting and evaluation* | X | - | - | - | - | - |
| Randomize | X | - | - | - | - | - |
| Order study lenses | X | - | - | - | - | - |

| Visit 1 Screening / Trial Lens Fitting and Evaluation | Visit 2 Baseline / Dispense Lens 1 | Visit 3 Week 1 Follow-up Lens 1 / Dispense Lens 2 | Visit 4 Week 1 Follow-up Lens 2 / Exit | Unscheduled<br>Visit | Early<br>Exit |
|---|---|---|---|---|---|
| | 4 -2/+2 days after Visit 1 | 8 -0/+3 days after Visit 2 | 8 -0/+3 days after Visit 3 | N/A | N/A |
| - | X | X | - | (X) | - |
| - | X | X | - | - | - |
| - | X | X (lens 1 and 2) | X | (X) | X |
| | Lens Fitting and Evaluation | Lens Fitting and Evaluation Dispense Lens 1 4 -2/+2 days after Visit 1 X X | Lens Fitting and Evaluation Dispense Lens 1 Lens 1 / Dispense Lens 2 4 -2/+2 days after Visit 1 8 -0/+3 days after Visit 2 X X X | Lens Fitting and Evaluation Dispense Lens 1 Lens 1 / Dispense Lens 2 / Exit Lens 2 / Exit 4 -2/+2 days after Visit 1 8 -0/+3 days after Visit 2 8 -0/+3 days after Visit 3 - X X - X - X X X | Lens Fitting and Evaluation Dispense Lens 1 Lens 1 / Dispense Lens 2 Lens 2 / Exit Lens 2 / Exit A -2/+2 days after Visit 1 X X X - X X X - X X - X X |

Document ID: V-CLN-0010097

| Procedure / Assessment | Visit 1 Screening / Trial Lens Fitting and Evaluation | Visit 2 Baseline / Dispense Lens 1 | Visit 3 Week 1 Follow-up Lens 1 / Dispense Lens 2 | Visit 4 Week 1 Follow-up Lens 2 / Exit | Unscheduled<br>Visit | Early<br>Exit |
|---|---|---|---|---|---|---|
| | | 4 -2/+2 days after Visit 1 | 8 -0/+3 days after Visit 2 | 8 -0/+3 days after Visit 3 | N/A | N/A |

| AEs | X | X | X | X | (X) | X |
|---------------------|---|---|---|---|-----|---|
| Device Deficiencies | X | X | X | X | (X) | X |
| Exit Form | - | - | - | X | - | X |

(X) assessment performed as necessary, e.g., decrease of VA by 2 lines or more with investigational product (IP)

<sup>\*</sup> Source only

 $<sup>\</sup>infty$  All ocular and targeted systemic medications/ medical history

